CLINICAL TRIAL: NCT06258057
Title: Safety of Tetanus, Diphtheria, Acellular Pertussis With 5 Acellular Pertussis Components (Tdap5) Vaccination During Pregnancy: A Cohort Study Using US Electronic Medical Record Data
Brief Title: Safety of Tetanus, Diphtheria, Acellular Pertussis With 5 Acellular Pertussis Components (Tdap5) Vaccination During Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: TD500066; U1111-1290-9165 (Registry Identifier: ICTRP); TD500066 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-01-12; First posted 2024-02-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pertussis (Whooping Cough)
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adacel-Exposed Cohort: Cohort will include all pregnant individuals with a record of Adacel vaccination during the third trimester of pregnancy (ie, first day of 27th week of gestation up to the end of pregnancy) and their offspring
  Interventions: Other: Not applicable / database analysis
- Tdap-Unvaccinated Comparator Cohort: Cohort will include all pregnant individuals meeting eligibility criteria and with no record of any Tdap vaccination from pregnancy onset date until the end of pregnancy and their offspring
  Interventions: Other: Not applicable / database analysis

INTERVENTIONS:
Other: Not applicable / database analysis — Not applicable / database analysis

SUMMARY:
The purpose of this study is to evaluate the safety of Adacel vaccine among pregnant individuals exposed to Adacel at any point between the 1st day of the 27th week of gestation up to the end of pregnancy and their offspring (ie, Adacel-exposed cohort), in comparison with pregnant individuals not vaccinated with any Tdap vaccines during pregnancy and their offspring (ie, Tdap-unvaccinated comparator cohort).

The primary objectives are to estimate incidence rates and relative risks for each prespecified pregnancy outcome in Adacel-exposed and Tdap-unvaccinated comparator cohorts and for each prespecified adverse birth outcome in the offspring of both cohorts.

The secondary objectives are to estimate incidence rates and relative risks for each prespecified adverse fetal and neonatal outcome in the offspring of Adacel-exposed and Tdap unvaccinated comparator cohorts and for each prespecified adverse outcome for pregnant individuals in both cohorts.

DETAILED DESCRIPTION:
Study outcomes to be assessed in electronic medical records between January 2016 to December 2025.

ELIGIBILITY:
Inclusion Criteria:

* For pregnant individuals:

  * Continuous enrollment, with no more than a 1-month administrative gap from 90 days prior to their last menstrual period (LMP)
  * Continuous enrollment for the duration of their pregnancy through delivery or termination of pregnancy (or 6 weeks postpartum for preeclampsia/eclampsia and 28 days for PPH) unless censored at death in order to capture study outcomes
  * At least 1 prenatal visit prior to 27 weeks of gestation during pregnancy
* For offspring:

  * Infants delivered by pregnant individuals who meet all the inclusion criteria above
  * With gestational age as calculated based on date of birth recorded in the EMR

Exclusion Criteria:

* For pregnant individuals:

  * Loss of pregnancy or with delivery before 27 weeks of gestation
  * Vaccinated with Boostrix® (Tdap vaccine, GSK), or with an unknown brand of Tdap vaccine, or Td (tetanus, diphtheria) vaccine during pregnancy
  * Vaccinated with any Tdap vaccine prior to the ACIP recommended optimal timeframe of ≥ 270/7 weeks of gestation
  * Received more than one Tdap vaccine during pregnancy
  * Vaccinated with one or more live vaccines during pregnancy
  * Pregnant individuals with multiple gestation pregnancies (eg, twins, triplets)
* For offspring:

  * Infants delivered by pregnant individuals who meet any of the exclusion criteria above

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant individuals and their offspring
Study Population: The study population will be comprised of 2 cohorts of pregnant individuals with pregnancy onset from 01 January 2016 through 31 December 2024. Infants born from this study population of pregnant individuals with singleton gestation pregnancies will be eligible for inclusion in this study. Eligible live born infants must be born on 01 October 2025 or prior to this date, to allow adequate follow-up time
Sampling Method: Non-Probability Sample
Enrollment: 365000 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome: Live birth | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of live births in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Pregnancy outcome: Still birth/fetal demise | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of still birth/fetal demise in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Pregnancy outcome: Therapeutic abortion | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of therapeutic abortion in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Birth outcome: Preterm birth | From 1st day of the 27th week of gestation and less than 37 weeks gestation
  Incidence rates of preterm birth in live born infants of both Adacel-exposed and Tdap-unvaccinated comparator cohorts
Birth outcome: Low birth weight | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of low birth weight in live born infants of both Adacel-exposed and Tdap-unvaccinated comparator cohorts
Birth outcome: Small for gestational age | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of small for gestational age in live born infants of both Adacel-exposed and Tdap-unvaccinated comparator cohorts

SECONDARY OUTCOMES:
Adverse neonatal outcome: Neonatal death | From birth up to 28 days post-birth
  Incidence rates of neonatal death in the offspring of Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse neonatal outcome: Neonatal sepsis | From birth up to 28 days post-birth
  Incidence rates of neonatal sepsis in the offspring of Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse neonatal outcome: Neonatal respiratory distress | From birth up to 28 days post-birth
  Incidence rates of neonatal respiratory distress in the offspring of Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse neonatal outcome: Congenital anomalies | From birth up to 28 days post-birth
  Incidence rates of congenital anomalies (major and minor) in the offspring of Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse neonatal outcome: Neonatal/early infancy intensive care admissions for bronchopulmonary dysplasia | From birth up to 28 days post-birth
  Incidence rates of neonatal/early infancy intensive care admissions for bronchopulmonary dysplasia in the offspring of Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse fetal outcome: Fetal growth arrest (restriction) | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of fetal growth arrest (restriction) in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Preterm labor | From 1st day of the 27th week of gestation and less than 37 weeks gestation
  Incidence rates of Preterm labor in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Preeclampsia/eclampsia | From 1st day of the 27th week of gestation up to 42 days postpartum
  Incidence rates of preeclampsia/eclampsia in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Postpartum hemorrhage | Within 24 hours of delivery up to 28 days postpartum
  Incidence rates of postpartum hemorrhage in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Placental abruption | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of placental abruption in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Premature rupture of membranes | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of premature rupture of membranes in Adacel-exposed and Tdap-unvaccinated comparator cohorts
Adverse outcomes in pregnant individuals: Chorioamnionitis | From 1st day of the 27th week of gestation up to 42 weeks gestation
  Incidence rates of chorioamnionitis in Adacel-exposed and Tdap-unvaccinated comparator cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org